CLINICAL TRIAL: NCT07002021
Title: Effectiveness Evaluation of the "Mosquito-Free Campus" Initiative on Dengue Fever Prevention and Control: A Cluster Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lin Xu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SunYat-senU20250516
Record Dates: First submitted 2025-05-25; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Dengue; Infection Prevention
Keywords: health education; schools; China
MeSH Terms: conditions — Dengue; Health Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive a health education intervention focused on dengue prevention every semester for 6 months
  Interventions: Combination Product: Health education
- No Intervention: Control (No Intervention): The control group will continue with their routine school health education for 6 months.

INTERVENTIONS:
Combination Product: Health education — The intervention group will receive a health education intervention focused on dengue prevention and campus environmental governance, while the control group will continue with their standard school health education without any additional intervention. An health education including the knowledge of dengue fever, harm of mosquitoes, and measures of mosquito control, will be developed and reviewed by an expert group. The campus environmental governance includes organizing campus environmental cleaning once a week, focusing on removing mosquito breeding places such as water containers.
  Arms: Intervention

SUMMARY:
The goal of this cluster randomized controlled trial is to evaluate the effect of health education interventions on the score of the knowledge, attitudes, and practices (KAP) of dengue in in primary and middle school students in the city of Guangzhou and Foshan in China.

Individuals aged 6 to 15 years who are in grades 1-9 in primary schools in Guangzhou and Foshan will be enrolled. 20 primary schools will be randomly selected, with half designated as intervention group schools and the remaining half as control group schools. The intervention group will receive a health education intervention focused on dengue prevention every semester for 6 months, while the control group will continue with their routine school health education for 6 months.

Researchers will compare the differences in the score of the KAP of dengue between the intervention and control groups after 6 months to see if health education can improve knowledge, attitudes and practices of dengue among primary and middle school students.

DETAILED DESCRIPTION:
Introduction: Dengue is one of the fastest spreading mosquito-borne infectious diseases in the world. Guangdong, as the core epidemic area of dengue fever in China, has experienced many large outbreaks of dengue in history due to its warm and humid climate, dense urbanization, and frequent communication with Southeast Asia. However, prevention and control measures in schools remains suboptimal. This study aims to improve the knowledge, attitudes, and practices (KAP) of dengue prevention and control among students, and reduce the density of mosquito vectors and the risk of dengue transmission in primary and middle schools.

Methods and analysis: This cluster randomized controlled trial will enroll 3940 students from 20 primary and middle schools in Guangzhou and Foshan City, China. Schools will be randomized to an intervention group receiving dengue health education and environmental governance or a control group receiving routine health education. The primary outcome is scores of KAP of students. Secondary outcomes include environmental mosquito vector index. Data will be collected through questionnaires, campus environment inspection, and self-reports at baseline and study conclusion.

Ethics and dissemination: Ethical approval has been sought from the Ethics Committee of the School of Public Health, Sun Yat-sen University. Findings from the study will be made accessible to key stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* Primary and middle school students within the age range of 6-15 years.
* The primary and middle schools are located in Yuexiu District, Baiyun District of Guangzhou city or Nanhai District of Foshan City.
* The schools have the necessary infrastructure, management level and resource allocation to participate in dengue fever prevention and control.
* The schools agree to implement the intervention measures during the research period.
* The schools are willing to provide baseline data and participate in subsequent assessments before the intervention is implemented.

Exclusion Criteria:

* Unwilling to participate in the project.
* Participants (students or staff members) are unable to participate in the intervention or withdraw from the study due to personal reasons.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3940 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
scores of the knowledge, attitudes, and practices (KAP) of dengue | From enrollment to the end of intervention in 6 months
  Regarding the knowledge, attitudes, and practices of dengue, each correct answer for the health literacy research questionnaire will be scored as one point, with incorrect answers receiving no points.

SECONDARY OUTCOMES:
mosquito vector index | From enrollment to the end of intervention in 6 months
  The mosquito vector index will be calculated as the number of mosquitoes captured in a fixed area divided by the total area.

IPD SHARING:
Plan to Share IPD: No